CLINICAL TRIAL: NCT00077870
Title: A Randomized, Placebo-Controlled, Multicenter, Blinded Phase I/II Study of the Safety of Escalating Doses of Ocrelizumab (PRO70769) in Subjects With Moderate to Severe Rheumatoid Arthritis Receiving Stable Doses of Concomitant Methotrexate
Brief Title: A Study to Evaluate the Safety of Escalating Doses of Ocrelizumab in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: ACT2847g
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Moderate to severe rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ocrelizumab

INTERVENTIONS:
Drug: ocrelizumab

SUMMARY:
This is a randomized, placebo-controlled, multicenter, blinded Phase I/II, investigator and subject-blinded study of the safety of escalating doses of ocrelizumab in combination with MTX in subjects with moderate to severe RA

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent and to comply with the requirements of the protocol
* Diagnosis of RA for at least 6 months according to the revised 1987 ACR criteria for the classification of RA
* Positive serum RF
* Current treatment for RA on an outpatient basis
* Contact your local site that is listed for more inclusion criteria

Exclusion Criteria:

* Bone or joint surgery (including joint fusion) within 8 weeks prior to screening or joint surgery planned within 24 weeks after randomization
* Rheumatic autoimmune disease other than RA or significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis, or Felty�s syndrome)
* Functional Class IV as defined by the ACR classification of functional status in RA
* History of or current inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) or other systemic rheumatic disorders (e.g., systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, overlap syndrome)
* Contact your local site that is listed for more exclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237
Dates: Start 2004-02; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ocrelizumab in subjects with moderate to severe RA

SECONDARY OUTCOMES:
Pharmacokinetics of ocrelizumab
Pharmacodynamics of ocrelizumab
Percentage of subjects with clinical responses according to American College of Rheumatology (ACR) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dummer, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Result] Genovese MC, Kaine JL, Lowenstein MB, Del Giudice J, Baldassare A, Schechtman J, Fudman E, Kohen M, Gujrathi S, Trapp RG, Sweiss NJ, Spaniolo G, Dummer W; ACTION Study Group. Ocrelizumab, a humanized anti-CD20 monoclonal antibody, in the treatment of patients with rheumatoid arthritis: a phase I/II randomized, blinded, placebo-controlled, dose-ranging study. Arthritis Rheum. 2008 Sep;58(9):2652-61. doi: 10.1002/art.23732. PMID 18759293